CLINICAL TRIAL: NCT02379000
Title: Transpupillary Thermotherapy (TTT) Alone Versus the Combined Therapy Consisting of TTT and Intravitreal Injection of Triamcinolone to Decrease Exudation in Choroidal Melanoma After Proton Beam Therapy
Brief Title: TTT Versus TTT and Triamcinolone to Decrease Exudation in Choroidal Melanoma After Proton Beam Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Dr. Ira Seibel, TTT Versus TTT and Triamcinolone to Decrease Exudation in Choroidal Melanoma After Proton Beam Therapy, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2404
Record Dates: First submitted 2015-02-23; First posted 2015-03-04 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Exudative Retinal Detachment; Uveal Melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transpupillary therapy alone (Active Comparator): Transpupillary thermotherapy is performed as monotherapy. It is performed with an infrared diode laser adapted to a slit-lamp biomicroscope at a wavelength of 810 nm and beam diameters of 0.5, 0.8, 1.2, 2.0, or 3.0 mm using a contact lens and through a dilated pupil. Each TTT spot was applied for a duration of about 1 minute to achieve a grayish-white color on the surface of the tumor. TTT could be repeated at intervals of 6-8 weeks with the goal of achieving a complete resolution of fluid
  Interventions: Procedure: Transpupillary thermotherapy
- TTT+Triamcinolone Acetonide (Active Comparator): transpupillary thermotherapy followed by an intravitreal injection of triamcinolone. It is performed with an infrared diode laser adapted to a slit-lamp biomicroscope at a wavelength of 810 nm and beam diameters of 0.5, 0.8, 1.2, 2.0, or 3.0 mm using a contact lens and through a dilated pupil. Each TTT spot was applied for a duration of about 1 minute to achieve a grayish-white color on the surface of the tumor. After an intravitreal injection of triamcinolone was perfomed under sterile conditions. TTT and triamcinolone injection could be repeated at intervals of 6-8 weeks with the goal of achieving a complete resolution of fluid.
  Interventions: Drug: Triamcinolone Acetonide; Procedure: Transpupillary thermotherapy

INTERVENTIONS:
Drug: Triamcinolone Acetonide — Under sterile conditions an intravitreal injection of trimcinolone acetonide 4 mg was performed.
  Other Names: Volon A
  Arms: TTT+Triamcinolone Acetonide
Procedure: Transpupillary thermotherapy — We delivered TTT with an infrared diode laser adapted to a slit-lamp biomicroscope at a wavelength of 810 nm and beam diameters of 0.5, 0.8, 1.2, 2.0, or 3.0 mm using a contact lens and through a dilated pupil. Each TTT spot was applied for a duration of about 1 minute to achieve a grayish-white color on the surface of the tumor.
  Other Names: TTT

SUMMARY:
Proton beam therapy is a safe irradiation modality for choroidal melanoma. But often after irradiation the exudation increases resulting in an exudative retinal detachment requiring vitreoretinal surgery. It is known that intravitreally injected triamcinolone and TTT is capable to decrease the exudation. If there is any advantage in a combined treatment this study will investigate.

DETAILED DESCRIPTION:
Proton beam therapy is an eye preserving irradiation modality for uveal melanoma. After proton beam therapy tumor related lipid exudation and exudative retinal detachment often increase. Therefore vitreoretinal surgery is sometimes required to reattach the retina to protect visual acuity. It is known that intravitreally injected triamcinolone and TTT is capable to decrease exudation. If there is any advantage in a combined treatment and if it is that effective to possibly avoid vitreoretinal surgery this study will investigate.

ELIGIBILITY:
Inclusion Criteria:

•exudation (tumor associated exudation/exudative retinal detachment) after proton beam therapy in choroidal melanoma and/or ciliary body melanoma

Exclusion criteria:

* Tumor recurrence
* Endoresection and / or previous vitrectomy
* Treatment with anti-angiogenic drugs or intravitreal corticosteroids or any other investigational drug within 3 months prior to randomisation
* Prior laser photocoagulation treatment within 3 months (focal / grid laser) or 6 months (panretinal) prior to study entry
* Known hypersensitivity against local anaesthetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Decrease of exudation, as indicated by compairing the extent of exudation measured in quadrants in color fundus photographs, autofluorescence imaging, and/or optical coherence tomogaphy. | 6 weeks, 6 months

SECONDARY OUTCOMES:
Toxic tumor syndrone and required secondary vitrectomy | 3 years
  If tumor relaxed lipid exudates or a neovascular glaucoma develop a secondary vitrectomy will be required to preserve the globe.

CONTACTS AND LOCATIONS:
Overall Officials: Ira Seibel, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] Desjardins L, Lumbroso-Le Rouic L, Levy-Gabriel C, Dendale R, Delacroix S, Nauraye C, Esteve M, Plancher C, Asselain B. Combined proton beam radiotherapy and transpupillary thermotherapy for large uveal melanomas: a randomized study of 151 patients. Ophthalmic Res. 2006;38(5):255-60. doi: 10.1159/000094834. Epub 2006 Jul 28. PMID 16888407
- [Background] Parrozzani R, Pilotto E, Dario A, Miglionico G, Midena E. Intravitreal triamcinolone versus intravitreal bevacizumab in the treatment of exudative retinal detachment secondary to posterior uveal melanoma. Am J Ophthalmol. 2013 Jan;155(1):127-133.e2. doi: 10.1016/j.ajo.2012.06.026. Epub 2012 Sep 18. PMID 22995029
- [Background] Seibel I, Cordini D, Willerding G, Riechardt AI, Joussen AM. Endodrainage, Tumor Photocoagulation, and Silicone Oil Tamponade for Primary Exudative Retinal Detachment due to Choroidal Melanoma Persisting after Proton Beam Therapy. Ocul Oncol Pathol. 2014 Oct;1(1):24-33. doi: 10.1159/000365333. Epub 2014 Jul 22. PMID 27175359